CLINICAL TRIAL: NCT04264741
Title: Transcranial Magnetic Stimulation for Treating Patients Under Methadone Maintenance Therapy Combined With Methamphetamine Abuse
Brief Title: Transcranial Magnetic Stimulation for Methadone Maintenance Therapy Combined With Methamphetamine Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HFJiang-004
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Methamphetamine Abuse
Keywords: repetitive transcranial magnetic stimulation (rTMS); methamphetamine abuse; methadone maintenance therapy; urine test; relapse
MeSH Terms: conditions — Recurrence | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS treatment group (Experimental): For rTMS treatment, we will stimulate the dorsal lateral prefrontal cortex of each patients using the iTBS pattern everyday. Treatment will lasted for 4 weeks.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- sham rTMS treatment group (Sham Comparator): For sham rTMS treatment, we will stimulate the dorsal lateral prefrontal cortex of each patients using the sham iTBS pattern and sham coil everyday. Treatment will lasted for 4 weeks.
  Interventions: Device: sham repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — The iTBS group received 900 pulses per day: 3-pulse 50-Hz bursts given every 200 ms (at 5 Hz), 2 s on and 8 s off for 5 min, at 100% resting motor threshold (rMT), over the left DLPFC (F3, EEG system) (4 weeks, 20 daily sessions). A figure-8-shaped Cool-B70 stimulation coil from MagPro X100 device (MagVenture, Farum, Denmark) was used for accurately targeted stimulation. Motor threshold was determined over the left motor cortex, by finding the lowest intensity that produced a motor response in the right abductor pollicis brevis muscles (APB), which produced five motor-evoked potentials responses of at least 50 mV in 10 trials.
  Arms: rTMS treatment group
Device: sham repetitive transcranial magnetic stimulation (rTMS) — The iTBS group received 900 pulses per day: 3-pulse 50-Hz bursts given every 200 ms (at 5 Hz), 2 s on and 8 s off for 5 min, at 100% resting motor threshold (rMT), over the left DLPFC (F3, EEG system) (4 weeks, 20 daily sessions). A figure-8-shaped sham Cool-B70 stimulation coil from MagPro X100 device (MagVenture, Farum, Denmark) was used for accurately targeted stimulation. Motor threshold was determined over the left motor cortex, by finding the lowest intensity that produced a motor response in the right abductor pollicis brevis muscles (APB), which produced five motor-evoked potentials responses of at least 50 mV in 10 trials.
  Arms: sham rTMS treatment group

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) has been used to treat opioid and methamphetamine addiction in previous studies, while no evidence was proved for patients methadone maintenance therapy with methamphetamine abuse. The aim of this study is to evaluating the effectiveness and safety of rTMS treatment for methamphetamine abuse in patients with methadone maintenance therapy.

DETAILED DESCRIPTION:
First, a multicenter, double-blind, randomized control study is going to be carried out. 60 recruited patients will be randomized assigned to the intervention group (40) and the control group (20), receiving either 4-week of repetitive transcranial magnetic stimulation (rTMS) treatment or 4-week of sham rTMS treatment. Both groups will receive 16-week urine drug test (1 time per week, 4 weeks before rTMS, 4 weeks during rTMS and 8 weeks after rTMS). Self-report methamphetamine use or urine test is set as primary outcome. Cognitive function and craving are also evaluated before and after the intervention. Functional magnetic resonance imaging (fMRI) is applied to investigate the potential neurobiological mechanism of rTMS treatment. This study will be very helpful to develop an evidence-based rTMS treatment protocols for methadone maintenance therapy with methamphetamine abuse and decrease risk of relapse for both the patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* Currently in methadone maintenance therapy
* In accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) for methamphetamine (MA) use disorders
* Junior high school degree or above
* Normal vision and hearing

Exclusion Criteria:

* Have a disease that affect cognitive function such as history of head injury, cerebrovascular disease, epilepsy, etc
* Have cognitive-promoting drugs in the last 6 months
* Other substance abuse or dependence in recent five years (except nicotine)
* Mental impairment, Intelligence Quotient (IQ) < 70
* Mental disorders according to DSM-5 criteria
* Physical diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Self-report drug use and urine test | 16 weeks
  Patients will be asked to report their drug use for 16 weeks every day and do urine tests once a week for 16 weeks. Loss of visit or rejecting to report or rejecting to do urine tests will be treated as drug use positive (relapse).

SECONDARY OUTCOMES:
Change of Craving assessed by Visual Analog Scale | 12 weeks
  Evaluate all participants' craving for for methamphetamine assessed by Visual Analog Scales (VAS). Score of VAS range from 0 to 10, and higher values represent high level of craving.
Cognitive function assessed by Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 12 weeks
  Evaluate all participants' cognitive function by Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Chinese version
Functional magnetic resonance imaging | 4 weeks
  Functional magnetic resonance imaging is collected once before and once after intervention, mainly collecting structural images, resting state, and task-based fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Jiang, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Wuhan Mental Health Center, Wuhan, China